CLINICAL TRIAL: NCT00195676
Title: A Multicenter Open-Label Continuation Study in Moderate to Severe Chronic Plaque Psoriasis Subjects Who Completed a Preceding Psoriasis Clinical Study With Adalimumab
Brief Title: Efficacy and Safety of Adalimumab in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Martin M. Okun, MD, PhD/Medical Director, Immunology, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M03-658; 2005-000095-41 (EudraCT Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2010-11-19 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

ARMS (1):
- Adalimumab (Other)
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — 40 mg every other week or 40 mg every week by subcutaneous injection
  Other Names: ABT-D2E7; Humira

SUMMARY:
The two objectives of this study were to evaluate long-term efficacy and safety of adalimumab treatment in participants who had moderate to severe chronic plaque psoriasis and to evaluate the effectiveness of adalimumab retreatment in participants who had therapeutic response to adalimumab and were then withdrawn from adalimumab treatment.

DETAILED DESCRIPTION:
Study M03-658 was a continuation study for participants with moderate to severe psoriasis who had participated in a prior psoriasis adalimumab study. Study M03-658 consisted of three sequential treatment periods. The first period was Period O, in which participants received open-label treatment with adalimumab (40 mg every other week or 40 mg every week) for a minimum of 104 weeks and a maximum of 252 weeks. Period O was the only period of the study until May 2008, when the subsequent periods were added via amendment to the protocol. At that time, participants who had achieved satisfactory therapeutic response (a Physician's Global Assessment [PGA] of 0, 1, or 2 [clear, minimal, or mild]) were given the opportunity to discontinue from the study or to continue and participate in the subsequent two periods. The second period was Period W, a maximum of 52 weeks, in which participants with a PGA of 2 (mild) or less were withdrawn from adalimumab treatment (i.e., participants received no treatment) until relapse of their psoriasis occurred (defined as a PGA of 3 [moderate] or worse). The third period was Period R, a 16-week period in which participants were retreated with open-label adalimumab (80 mg initial dose followed by 40 mg every other week). Period O was designed to evaluate the first objective regarding long-term efficacy and safety of adalimumab treatment, and Period R was designed to evaluate the effectiveness of adalimumab retreatment following relapse. Specific subsets of the study population that were identified as the populations of interest were the modified intent-to-treat populations for Period W and Period R, and these are described further in the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Subject was age 18 or older and in good health (Investigator discretion) with a recent stable medical history.
* Subjects who met the requirements from previous adalimumab psoriasis study participation.

Exclusion Criteria:

* Subject considered by the Investigator, for any reason, to be an unsuitable candidate for the study.
* Female subject who was pregnant or breast-feeding or considering becoming pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1469 (Actual)
Dates: Start 2004-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Okun, MD, PhD, Study Director — Abbott
Locations (104):
- United States (66):
  - Site Reference ID/Investigator# 1263, Birmingham, Alabama
  - Site Reference ID/Investigator# 1259, Buckner 13075 PI, Alabama
  - Site Reference ID/Investigator# 2427, Scottsdale, Arizona
  - Site Reference ID/Investigator# 2433, Tucson, Arizona
  - Site Reference ID/Investigator# 100, Little Rock, Arkansas
  - Site Reference ID/Investigator# 1798, Bakersfield, California
  - Site Reference ID/Investigator# 122, Fresno, California
  - Site Reference ID/Investigator# 1669, Irvine, California
  - Site Reference ID/Investigator# 1285, Oceanside, California
  - Site Reference ID/Investigator# 86, San Diego, California
  - Site Reference ID/Investigator# 1679, Santa Monica, California
  - Site Reference ID/Investigator# 1677, Torrance, California
  - Site Reference ID/Investigator# 1269, Longmont, Colorado
  - Site Reference ID/Investigator# 1275, New Haven, Connecticut
  - Site Reference ID/Investigator# 96, Jacksonville, Florida
  - Site Reference ID/Investigator# 2431, Pinellas Park, Florida
  - Site Reference ID/Investigator# 1273, South Miami, Florida
  - Site Reference ID/Investigator# 2432, West Palm Beach, Florida
  - Site Reference ID/Investigator# 98, Alpharetta, Georgia
  - Site Reference ID/Investigator# 1674, Newnan, Georgia
  - Site Reference ID/Investigator# 1670, Snellville, Georgia
  - Site Reference ID/Investigator# 1264, Chicago, Illinois
  - Site Reference ID/Investigator# 1801, Maywood, Illinois
  - Site Reference ID/Investigator# 1681, Springfield, Illinois
  - Site Reference ID/Investigator# 1267, Indianapolis, Indiana
  - Site Reference ID/Investigator# 1671, Indianapolis, Indiana
  - Site Reference ID/Investigator# 1258, Louisville, Kentucky
  - Site Reference ID/Investigator# 1281, Shreveport, Louisiana
  - Site Reference ID/Investigator# 1668, Andover, Massachusetts
  - Site Reference ID/Investigator# 1683, Boston, Massachusetts
  - Site Reference ID/Investigator# 83, Worcester, Massachusetts
  - Site Reference ID/Investigator# 93, Ann Arbor, Michigan
  - Site Reference ID/Investigator# 92, Fridley, Minnesota
  - Site Reference ID/Investigator# 1262, Minneapolis, Minnesota
  - Site Reference ID/Investigator# 1657, St Louis, Missouri
  - Site Reference ID/Investigator# 89, St Louis, Missouri
  - Site Reference ID/Investigator# 1673, Omaha, Nebraska
  - Site Reference ID/Investigator# 2119, New Brunswick, New Jersey
  - Site Reference ID/Investigator# 1672, New York, New York
  - Site Reference ID/Investigator# 1797, New York, New York
  - Site Reference ID/Investigator# 95, New York, New York
  - Site Reference ID/Investigator# 1655, New York, New York
  - Site Reference ID/Investigator# 88, Rochester, New York
  - Site Reference ID/Investigator# 1256, Williamsville, New York
  - Site Reference ID/Investigator# 1266, Raleigh, North Carolina
  - Site Reference ID/Investigator# 1265, Cincinnati, Ohio
  - Site Reference ID/Investigator# 90, Cleveland, Ohio
  - Site Reference ID/Investigator# 2434, Columbus, Ohio
  - Site Reference ID/Investigator# 1260, Lake Oswego, Oregon
  - Site Reference ID/Investigator# 1667, Portland, Oregon
  - Site Reference ID/Investigator# 121, Portland, Oregon
  - Site Reference ID/Investigator# 1323, Hershey, Pennsylvania
  - Site Reference ID/Investigator# 1277, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 99, Johnston, Rhode Island
  - Site Reference ID/Investigator# 1676, Providence, Rhode Island
  - Site Reference ID/Investigator# 97, Greer, South Carolina
  - Site Reference ID/Investigator# 5199, Mt. Pleasant, South Carolina
  - Site Reference ID/Investigator# 1800, Goodlettsville, Tennessee
  - Site Reference ID/Investigator# 1282, Nashville, Tennessee
  - Site Reference ID/Investigator# 87, Dallas, Texas
  - Site Reference ID/Investigator# 1279, Houston, Texas
  - Site Reference ID/Investigator# 1665, San Antonio, Texas
  - Site Reference ID/Investigator# 1268, Tyler, Texas
  - Site Reference ID/Investigator# 2079, Salt Lake City, Utah
  - Site Reference ID/Investigator# 123, Norfolk, Virginia
  - Site Reference ID/Investigator# 1653, Seattle, Washington
- Austria (3):
  - Site Reference ID/Investigator# 2181, Graz
  - Site Reference ID/Investigator# 2180, Innsbruck
  - Site Reference ID/Investigator# 2176, Vienna
- Belgium (2):
  - Site Reference ID/Investigator# 2554, Brussels
  - Site Reference ID/Investigator# 2179, Edegem
- Canada (17):
  - Site Reference ID/Investigator# 1629, Calgary, Alberta
  - Site Reference ID/Investigator#1641, Edmonton, Alberta
  - Site Reference ID/Investigator# 104, Vancouver, British Columbia
  - Site Reference ID/Investigator# 1635, St. John's, Newfoundland and Labrador
  - Site Reference ID/Investigator# 120, St. John's, Newfoundland and Labrador
  - Site Reference ID/Investigator# 94, Halifax, Nova Scotia
  - Site Reference ID/Investigator# 1640, Hamilton, Ontario
  - Site Reference ID/Investigator# 1636, London, Ontario
  - Site Reference ID/Investigator# 1639, North Bay, Ontario
  - Site Reference ID/Investigator# 1633, Toronto, Ontario
  - Site Reference ID/Investigator# 1631, Waterloo, Ontario
  - Site Reference ID/Investigator# 103, Windsor, Ontario
  - Site Reference ID/Investigator# 102, Montreal, Quebec
  - Site Reference ID/Investigator# 1637, Montreal, Quebec
  - Site Reference ID/Investigator# 101, Montreal, Quebec
  - Site Reference ID/Investigator# 1802, Québec, Quebec
  - Site Reference ID/Investigator# 1647, Westmount, Quebec
- France (4):
  - Site Reference ID/Investigator# 2553, Créteil
  - Site Reference ID/Investigator# 2191, Nice
  - Site Reference ID/Investigator# 2190, Paris
  - Site Reference ID/Investigator# 2189, Saint-Etienne
- Germany (4):
  - Site Reference ID/Investigator# 2198, Frankfurt
  - Site Reference ID/Investigator# 2543, Kiel
  - Site Reference ID/Investigator# 2188, Münster
  - Site Reference ID/Investigator# 2187, Tübingen
- Poland (2):
  - Site Reference ID/Investigator# 2178, Gdansk
  - Site Reference ID/Investigator# 2177, Płock
- Puerto Rico (2):
  - Site Reference ID/Investigator# 2194, Cagaus
  - Site Reference ID/Investigator# 5507, Carolina
- Spain (3):
  - Site Reference ID/Investigator# 2182, Madrid
  - Site Reference ID/Investigator# 2185, Seville
  - Site Reference ID/Investigator# 2183, Valencia
- Site Reference ID/Investigator# 2193, Geneva, Switzerland

REFERENCES:
- [Derived] Gordon K, Papp K, Poulin Y, Gu Y, Rozzo S, Sasso EH. Long-term efficacy and safety of adalimumab in patients with moderate to severe psoriasis treated continuously over 3 years: results from an open-label extension study for patients from REVEAL. J Am Acad Dermatol. 2012 Feb;66(2):241-51. doi: 10.1016/j.jaad.2010.12.005. Epub 2011 Jul 14. PMID 21752491
- [Derived] Papp K, Crowley J, Ortonne JP, Leu J, Okun M, Gupta SR, Gu Y, Langley RG. Adalimumab for moderate to severe chronic plaque psoriasis: efficacy and safety of retreatment and disease recurrence following withdrawal from therapy. Br J Dermatol. 2011 Feb;164(2):434-41. doi: 10.1111/j.1365-2133.2010.10139.x. PMID 21083543

RESULTS

PARTICIPANT FLOW:
Groups:
- All Adalimumab Treatment: All participants in the study who received at least one dose of adalimumab. In this study, participants were treated with adalimumab 40 mg every other week (eow) or 40 mg every week by subcutaneous injection (SC) in Period O and then were retreated with open-label adalimumab 40 mg eow SC (after an 80 mg initial dose) in Period R after withdrawal from adalimumab treatment in Period W.
Period: Period O - Open-label Treatment
Arm/Group | All Adalimumab Treatment
Started | 1468 (Number receiving adalimumab in Period O (1 additional participant enrolled but did not receive drug))
Completed | 862 (254 Period O completers did not consent or were not eligible to continue into Period W and Period R.)
Not Completed | 606
Not completed — Adverse Event | 82
Not completed — Death | 6
Not completed — Lack of Efficacy | 198
Not completed — Lost to Follow-up | 91
Not completed — Protocol Violation | 12
Not completed — Withdrawal by Subject | 147
Not completed — Administrative reasons | 2
Not completed — Other reasons | 68
Period: Period W (Withdrawal) - No Treatment
Arm/Group | All Adalimumab Treatment
Started | 608 (Period O completers with a Physician's Global Assessment =<2 who continued into Periods W and R.)
Completed | 0 (Non-completers may have entered Period R, whether or not they relapsed (PGA >= 3).)
Not Completed | 608
Not completed — Adverse Event | 4
Not completed — Death | 2
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 46
Not completed — Relapse (PGA >= 3) | 397
Not completed — Period W Close-out | 129
Not completed — Administrative reasons | 1
Not completed — Other reasons | 18
Period: Period R - Retreatment 16 Weeks
Arm/Group | All Adalimumab Treatment
Started | 525 (Number who entered from Period W, including those who did and did not relapse in that period.)
Completed | 490
Not Completed | 35
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 5
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 9
Not completed — Other reasons | 6

BASELINE CHARACTERISTICS:
Arm/Group | All Adalimumab Treatment
Number analyzed (Participants) | 1468
Age Continuous [Mean (Standard Deviation); unit: years] | 44.1 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 470
  Male | 998
Region of Enrollment [Number; unit: participants]
  United States | 802
  Canada | 501
  Austria | 34
  Belgium | 15
  France | 45
  Switzerland | 3
  Spain | 20
  Poland | 12
  Germany | 36

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Percentage of Participants With a Physician's Global Assessment of Clear or Minimal at Week 60
Description: The Physician's Global Assessment [PGA] was scored by the physician using a 6-point scale (0-5) for the degree of overall lesion severity, where 0 = clear, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, and 5 = very severe. Subjects with a PGA of Clear or Minimal overall lesion severity had scores of 0 or 1.
Time Frame: Week 60
Population: A subset of the All Adalimumab Treatment population who initiated treatment with an adalimumab 40 mg every other week (eow) injection or placebo injection in a prior study. Results were analyzed using Last Observation Carried Forward (LOCF) imputation for missing values.
Measure: Number; unit: percentage of participants
Groups:
- Period O Adalimumab EOW Treatment Population: Participants in the All Adalimumab Treatment population who initiated treatment with an adalimumab 40 mg every other week (eow) injection or placebo injection in a prior study.
Arm/Group | Period O Adalimumab EOW Treatment Population
Number analyzed (Participants) | 1256
percentage of participants | 50.6

2. Other Pre Specified Outcome: Percentage of Participants With a Physician's Global Assessment of Clear or Minimal at Week 120
Description: as for outcome 1
Time Frame: Week 120
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Period O Adalimumab EOW Treatment Population
Number analyzed (Participants) | 1256
percentage of participants | 46.3

3. Primary Outcome: Percentage of Participants With a Physician's Global Assessment of Clear or Minimal at Week 16 of Period R
Description: as for outcome 1
Time Frame: Week 16 of Period R
Population: The Period R Modified Intent-to-Treat population included 178 participants who relapsed and 107 participants who did not relapse in Period W when therapy was withdrawn; all received Period R adalimumab 40 mg every other week (after an 80 mg initial dose). Results were analyzed using non-responder imputation (NRI) for missing values.
Measure: Number; unit: percentage of participants
Groups:
- Period R Modified Intent-to-Treat Population: Participants of the Period W Modified Intent-to-Treat(mITT) Population who received at least one retreatment dose of adalimumab 40 mg every other week in Period R. The Period W mITT Population had entered Period W from Period O with stable psoriasis control [i.e., had a PGA of 0 or 1 at the last 2 consecutive visits in Period O, at least 12 weeks apart, and were on adalimumab 40 mg every other week for the last 12 weeks of Period O).
Arm/Group | Period R Modified Intent-to-Treat Population
Number analyzed (Participants) | 285
percentage of participants | 76.5

4. Other Pre Specified Outcome: Percentage of Participants Who Achieved a Psoriasis Area and Severity Index 75 (PASI 75) Response at Week 60
Description: Psoriasis Area and Severity Index (PASI) scores were calculated from assessments at 4 designated anatomical sites (head, upper extremities, trunk, lower extremities) using both severity and area subscores (i.e., degree of and amount of psoriatic involvement per site). PASI scores range from 0.0 (best) to 72.0 (worst), with the highest score representing complete erythroderma of the severest degree. Positive percent decreases indicate improvement, with the best improvement being 100%. A PASI 75 response was at least a 75% reduction in PASI score from baseline PASI score of the initial study.
Time Frame: Week 60
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Period O Adalimumab EOW Treatment Population
Number analyzed (Participants) | 1256
percentage of participants | 61.4

5. Other Pre Specified Outcome: Percentage of Participants Who Achieved a Psoriasis Area and Severity Index 75 (PASI 75) Response at Week 120
Description: as for outcome 4
Time Frame: Week 120
Population: A subset of the the All Adalimumab Treatment population who initiated treatment with an adalimumab 40 mg every other week (eow) injection or placebo injection in a prior study. Results were analyzed using Last Observation Carried Forward (LOCF) imputation for missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Period O Adalimumab EOW Treatment Population
Number analyzed (Participants) | 1256
percentage of participants | 57.3

6. Other Pre Specified Outcome: Time to Relapse in Period W
Description: Relapse of psoriasis was defined as a Physician's Global Assessment (assessment of overall lesion severity) score of greater than or equal to 3 (3=moderate; 4=severe; 5=very severe).
Time Frame: Period W
Population: Participants in the Period W Modified Intent-to-Treat Population who had relapsed (defined by a PGA of greater than or equal to 3) during Period W and had at least one post-baseline PGA assessment in Period W.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Period W Modified Intent-to-treat Population: Participants from Period O who entered Period W with a PGA of 0 or 1 for the last 2 consecutive visits of Period O, at least 12 weeks apart, and received adalimumab 40 mg every other week for at least 12 weeks prior to entering Period W.
Arm/Group | Period W Modified Intent-to-treat Population
Number analyzed (Participants) | 339
days | 141 [127 to 146]

7. Other Pre Specified Outcome: Percentage of Period R Modified Intent-to-Treat Participants Who Relapsed in Period W and Subsequently Had a Physician's Global Assessment of Clear or Minimal at Week 16 of Period R
Description: as for outcome 1
Time Frame: Week 16 of Period R
Population: Participants in the Period R mITT population who had relapsed (had a PGA of greater than or equal to 3) with adalimumab treatment withdrawal during Period W. Results were analyzed using non-responder imputation (NRI) for missing values.
Measure: Number; unit: percentage of participants
Groups:
- Period R mITT Population Relapsed in Period W: A subset of the Period R modified Intent-to-Treat (mITT) population who had relapsed in Period W after adalimumab therapy was withdrawn.
Arm/Group | Period R mITT Population Relapsed in Period W
Number analyzed (Participants) | 178
percentage of participants | 69.1

8. Other Pre Specified Outcome: Percentage of Period R Modified Intent-to-Treat Participants Who Did Not Relapse in Period W and Subsequently Had a Physician's Global Assessment of Clear or Minimal at Week 16 of Period R
Description: as for outcome 1
Time Frame: Week 16 of Period R
Population: Participants in the Period R mITT population who did not relapse (did not have a PGA greater than or equal to 3) with adalimumab treatment withdrawal during Period W. Results were analyzed using non-responder imputation (NRI) for missing values.
Measure: Number; unit: percentage of participants
Groups:
- Period R Modified Intent-to-Treat Not Relapsed in Period W: A subset of the Period R modified Intent-to-Treat (mITT) population who had not relapsed (i.e., PGA not greater than or equal to 3) in Period W after adalimumab therapy was withdrawn.
Arm/Group | Period R Modified Intent-to-Treat Not Relapsed in Period W
Number analyzed (Participants) | 107
percentage of participants | 88.8

ADVERSE EVENTS:
Time Frame: 2,095 days(approximately 5.7 years), including adalimumab exposure in prior studies
Description: Adverse events reported from the start of adalimumab treatment until 70 days after discontinuation of adalimumab treatment were defined as treatment-emergent and are displayed.
Arm/Group | All Adalimumab Treatment
Serious Adverse Events (participants affected / at risk) | 189/1468
Other Adverse Events (participants affected / at risk) | 1036/1468
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Adalimumab Treatment (N=1468)
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 3
Arrhythmia (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 3
Cardiac tamponade (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 10
Coronary artery occlusion (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 5
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia paroxysmal (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Otosclerosis (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Abdominal adhesions (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Enterocele (Gastrointestinal disorders) | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Intra-abdominal haematoma (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal rupture (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 3
Salivary gland mass (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 2
Localised oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Colecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Abscess (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Appendicitis perforated (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 6
Disseminated tuberculosis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Epiglottitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis escherichia coli (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Haematoma infection (Infections and infestations) | 1
Hepatitis C (Infections and infestations) | 1
Human ehrlichiosis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 2
Meningitis viral (Infections and infestations) | 1
Necrotising pasciitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Paratyphoid fever (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia legionella (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Staphylococcal abscess (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Device failure (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 4
Postprocedural haemorrhage (Injury, poisoning and procedural complications) | 3
Procedural pain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 3
Central obesity (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Metabolic syndrome (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Agnosia (Nervous system disorders) | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1
Brain mass (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 1
Hypoxic encephalopathy (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paresis (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3
Alcohol withdrawal syndrome (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Bipolar I disorder (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Cyclothymic disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 4
Depression suicidal (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 5
Renal colic (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Vesicoureteric reflux (Renal and urinary disorders) | 1
Bartholinitis (Reproductive system and breast disorders) | 1
Breast enlargement (Reproductive system and breast disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Cystocele (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 4
Ovarian cyst (Reproductive system and breast disorders) | 1
Perineal fistula (Reproductive system and breast disorders) | 1
Rectocele (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Excessive skin (Skin and subcutaneous tissue disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Physical abuse (Social circumstances) | 1
Abortion induced (Surgical and medical procedures) | 3
Aortic aneurysm (Vascular disorders) | 2
Aortic stenosis (Vascular disorders) | 1
Arterial stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Venous insufficiency (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Adalimumab Treatment (N=1468)
Diarrhoea (Gastrointestinal disorders) | 83
Nausea (Gastrointestinal disorders) | 82
Injection site reaction (General disorders) | 74
Bronchitis (Infections and infestations) | 116
Influenza (Infections and infestations) | 113
Nasopharyngitis (Infections and infestations) | 391
Sinusitis (Infections and infestations) | 150
Upper respiratory tract infection (Infections and infestations) | 298
Muscle strain (Injury, poisoning and procedural complications) | 84
Arthralgia (Musculoskeletal and connective tissue disorders) | 156
Back pain (Musculoskeletal and connective tissue disorders) | 110
Pain in extremity (Musculoskeletal and connective tissue disorders) | 75
Headache (Nervous system disorders) | 164
Cough (Respiratory, thoracic and mediastinal disorders) | 94
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 81
Hypertension (Vascular disorders) | 163

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.